CLINICAL TRIAL: NCT02910466
Title: A Phase 4, Open-Label, Single-Center Clinical Study of Extended Use of rhPTH(1-84) in Hypoparathyroidism
Brief Title: A Study of Extended Use of Recombinant Human Parathyroid Hormone (rhPTH(1-84)) in Hypoparathyroidism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP634-402
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Results first posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Chronic Hypoparathyroidism; Hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- rhPTH(1-84) (Experimental): Participants will receive 25, 50, 75, and 100 microgram (mcg) of rhPTH(1-84) subcutaneous injection to the thigh via a multidose pen injector device once daily for 36 months. The dose will be individualized based on albumin-corrected serum calcium (ACSC) and 24-hour calcium urinary excretion to achieve a serum calcium level in the lower half of the normal range.
  Interventions: Drug: rhPTH(1-84)

INTERVENTIONS:
Drug: rhPTH(1-84) — Participants will receive 25, 50, 75, and 100 microgram (mcg) of rhPTH(1-84) subcutaneous injection to the thigh via a multidose pen injector device once daily for 36 months. The dose will be individualized based on Albumin-corrected Serum Calcium (ACSC) and 24-hour calcium urinary excretion to achieve a serum calcium level in the lower half of the normal range.

SUMMARY:
Chronic hypoparathyroidism is a life-long and irreversible disease for which the chronic administration of rhPTH(1-84) is a potential treatment option. The group of participants in the AAAE0544 core study has been taking rhPTH(1-84) for the treatment of hypoparathyroidism for up to 11 years. This study is designed to extend this experience and gain knowledge about how safe and effective rhPTH(1-84) is in participants with hypoparathyroidism over a long-term duration.

ELIGIBILITY:
Inclusion Criteria

* Participants that are currently or previously enrolled in the core study (AAAE0544 [NCT01199614]) and have maintained uninterrupted therapy with recombinant human parathyroid hormone (rhPTH(1-84)) (transient interruptions of up to 1 month continuously off treatment may be allowed).
* Signed and dated informed consent form (ICF).
* Adult men and women 18 to 85 years of age.
* History of hypoparathyroidism for at least 12 months prior to rhPTH(1-84) treatment, defined by the requirement for supplemental calcium and/or active vitamin D to maintain serum calcium along with an undetectable or insufficient Parathyroid hormone (PTH) concentration.
* Able to perform daily subcutaneous (SC) self-injections of study medication (or have designee perform injection).
* Willingness and ability to understand and comply with the protocol. Women must agree to pregnancy testing and acceptable methods of contraception, as detailed in the protocol.

Exclusion Criteria

* The participant is treated or has been treated with any investigational drug, aside from rhPTH(1-84), within 30 days of consent.
* As assessed by the investigator, the participant has any safety or medical issues that contraindicate participation in the study.
* The participant and/or the participant's parent(s) or legally-authorized representative(s) are unable to understand the nature, scope, and possible consequences of the study.
* The participant is unable to comply with the protocol, example, uncooperative with protocol schedule, refusal to agree to all of the study procedures, inability to return for evaluations, or is otherwise unlikely to complete the study, as determined by the investigator or the medical monitor.
* The participant is pregnant or lactating.
* Participants who are at increased baseline risk for osteosarcoma such as participant with Paget's disease of bone or unexplained new elevations of alkaline phosphatase, participants with hereditary disorders predisposing to osteosarcoma or participants with a prior history of external beam or implant radiation therapy involving the skeleton.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Ayodele O, Rejnmark L, Mu F, Lax A, Berman R, Swallow E, Gosmanova EO. Five-Year Estimated Glomerular Filtration Rate in Adults with Chronic Hypoparathyroidism Treated with rhPTH(1-84): A Retrospective Cohort Study. Adv Ther. 2022 Nov;39(11):5013-5024. doi: 10.1007/s12325-022-02292-1. Epub 2022 Aug 26. PMID 36018496
- [Derived] Rejnmark L, Ayodele O, Lax A, Mu F, Swallow E, Gosmanova EO. The risk of chronic kidney disease development in adult patients with chronic hypoparathyroidism treated with rhPTH(1-84): A retrospective cohort study. Clin Endocrinol (Oxf). 2023 Apr;98(4):496-504. doi: 10.1111/cen.14813. Epub 2022 Aug 28. PMID 35974422
- [Derived] Chen KS, Gosmanova EO, Curhan GC, Ketteler M, Rubin M, Swallow E, Zhao J, Wang J, Sherry N, Krasner A, Bilezikian JP. Five-year Estimated Glomerular Filtration Rate in Patients With Hypoparathyroidism Treated With and Without rhPTH(1-84). J Clin Endocrinol Metab. 2020 Oct 1;105(10):e3557-65. doi: 10.1210/clinem/dgaa490. PMID 32738041
- [Derived] Tay YD, Tabacco G, Cusano NE, Williams J, Omeragic B, Majeed R, Gomez Almonte M, Bilezikian JP, Rubin MR. Therapy of Hypoparathyroidism With rhPTH(1-84): A Prospective, 8-Year Investigation of Efficacy and Safety. J Clin Endocrinol Metab. 2019 Nov 1;104(11):5601-5610. doi: 10.1210/jc.2019-00893. PMID 31310310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single site in the United States between 27 October 2016 (first participant first visit) and 20 December 2019 (last participant last visit).
Pre-assignment Details: A total of 39 participants were enrolled in the study who were treated in the core AAAE0544 (NCT01199614) study, out of which, 36 participants received treatment in this study. This study reports the additional data only for the current study (SHP634-402) which is on long term safety and efficacy of over 36 months of exposure to rhPTH(1-84), and the results for core study AAAE0544 (NCT01199614) will be posted separately, as planned.
Groups:
- rhPTH(1-84): Participants received 25 micrograms (mcg) of rhPTH(1-84) with an upwards increments to 50, 75, and 100 mcg subcutaneous (SC) injection to the thigh via a multi-dose pen injector device once daily for 36 months of treatment period. The dose of rhPTH(1 84) was individualized based on albumin-corrected serum calcium (ACSC) and 24-hour calcium urinary excretion at investigator's discretion to achieve a serum calcium level in the lower half of the normal range (8 and 9 milligram/deciliter [mg/dL]).
Period: Overall Study
Arm/Group | rhPTH(1-84)
Started | 39
Safety Set (The safety population consisted of all enrolled participants who received at least 1 dose of rhPTH(1-84) regardless of study (SHP634-402 or AAAE0544 [NCT01199614] core study).) | 39
Treated | 36
Completed | 0
Not Completed | 39
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 5
Not completed — Due to Food and Drug Administration (FDA) recall | 29
Not completed — Participant didn't meet inclusion criteria | 1

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all enrolled participants who received at least 1 dose of rhPTH(1-84) regardless of study (SHP634-402 or AAAE0544 [NCT01199614] core study).
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.9 (12.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 38
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (402) in Concentration of Albumin-corrected Serum Calcium (ACSC) at Month 6
Description: Baseline (402) was defined as the last available pre-dose value in SHP634-402.
Time Frame: Baseline (402), Month 6
Population: Safety population consisted of all enrolled participants who received at least 1 dose of rhPTH(1-84) regardless of study (SHP634-402 or AAAE0544 [NCT01199614] core study). Here, overall number of participants analyzed refer to the participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Millimole per liter (mmol/L)
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 23
Millimole per liter (mmol/L) | -0.005 (0.1546)

2. Primary Outcome: Change From Baseline (402) in Concentration of Albumin-corrected Serum Calcium (ACSC) at Month 12
Description: Baseline (402) was defined as the last available pre-dose value in SHP634-402.
Time Frame: Baseline (402), Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 29
mmol/L | 0.069 (0.1838)

3. Primary Outcome: Change From Baseline (402) in Concentration of Albumin-corrected Serum Calcium (ACSC) at Month 18
Description: Baseline (402) was defined as the last available pre-dose value in SHP634-402.
Time Frame: Baseline (402), Month 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 30
mmol/L | 0.066 (0.2158)

4. Primary Outcome: Change From Baseline (402) in Concentration of Albumin-corrected Serum Calcium (ACSC) at Month 24
Description: Baseline (402) was defined as the last available pre-dose value in SHP634-402.
Time Frame: Baseline (402), Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 27
mmol/L | 0.112 (0.2314)

5. Primary Outcome: Change From Baseline (402) in Concentration of Albumin-corrected Serum Calcium (ACSC) at Month 30
Description: Baseline (402) was defined as the last available pre-dose value in SHP634-402.
Time Frame: Baseline (402), Month 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 21
mmol/L | 0.145 (0.2447)

6. Primary Outcome: Change From Baseline (402) in Concentration of Albumin-corrected Serum Calcium (ACSC) at Month 36
Description: Baseline (402) was defined as the last available pre-dose value in SHP634-402.
Time Frame: Baseline (402), Month 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 1
mmol/L | 0.170 (NA) — Standard deviation could not be calculated because single participant was analyzed.

7. Primary Outcome: Change From Baseline (402) in Concentration of Albumin-corrected Serum Calcium (ACSC) at End of Treatment (EOT) (up to Month 36)
Description: Baseline (402) was defined as the last available pre-dose value in SHP634-402. EOT was defined as the last determination of response during the treatment period (from the date of first dose to the date of last dose + 1 day), was analyzed in addition to the scheduled visits.
Time Frame: Baseline (402), EOT (up to Month 36)
Population: Safety population consisted of all enrolled participants who received at least 1 dose of rhPTH(1-84) regardless of study (SHP634-402 or AAAE0544 [NCT01199614] core study). Here, overall number of participants analyzed refer to the participants evaluable for this outcome measure. Due to the FDA recall, no participant received rhPTH for more than 36 months in the study.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 33
mmol/L | 0.135 (0.2260)

8. Secondary Outcome: Percentage of Participants Who Achieved ACSC Concentrations Above, Below, or in the Range of 1.875 mmol/L (7.5 Milligram Per Deciliter [mg/dL]) to Upper Limit of Normal (ULN) at Month 6, 12, 18, 24, 30, 36 and EOT (up to Month 36)
Description: EOT was defined as the last determination of response during the treatment period (from the date of first dose to the date of last dose + 1 day), was analyzed in addition to the scheduled visits. Albumin-corrected Serum Calcium (mmol/L) = Total Calcium (mmol/L) + 0.02 * (40 gram per liter [g/L] - Albumin [g/L]).
Time Frame: At Month 6, 12, 18, 24, 30, 36 and EOT (up to Month 36)
Population: Safety population: all enrolled participants who received at least 1 dose of rhPTH(1-84) regardless of study (SHP634-402 or AAAE0544 [NCT01199614] core study). Here, overall number of participants analyzed refer to the participants evaluable for this outcome measure and "number analyzed" refer to participants evaluable for this outcome at given categories. Due to the FDA recall, no participant received rhPTH for more than 36 months in the study.
Measure: Number; unit: Percentage of participants
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 36
Percentage of participants
  At Month 6: less than (<) 1.875 mmol/L: number analyzed (Participants) | 24
  At Month 6: less than (<) 1.875 mmol/L | 20.8
  At Month 6: 1.875 mmol/L to ULN: number analyzed (Participants) | 24
  At Month 6: 1.875 mmol/L to ULN | 79.2
  At Month 6: >ULN: number analyzed (Participants) | 24
  At Month 6: >ULN | 0
  At Month 12: <1.875 mmol/L: number analyzed (Participants) | 32
  At Month 12: <1.875 mmol/L | 31.3
  At Month 12: 1.875 mmol/L to ULN: number analyzed (Participants) | 32
  At Month 12: 1.875 mmol/L to ULN | 65.6
  At Month 12: > ULN: number analyzed (Participants) | 32
  At Month 12: > ULN | 3.1
  At Month 18: <1.875 mmol/L: number analyzed (Participants) | 33
  At Month 18: <1.875 mmol/L | 24.2
  At Month 18: 1.875 mmol/L to ULN: number analyzed (Participants) | 33
  At Month 18: 1.875 mmol/L to ULN | 75.8
  At Month 18: >ULN: number analyzed (Participants) | 33
  At Month 18: >ULN | 0
  At Month 24: <1.875 mmol/L: number analyzed (Participants) | 30
  At Month 24: <1.875 mmol/L | 16.7
  At Month 24: 1.875 mmol/L to ULN: number analyzed (Participants) | 30
  At Month 24: 1.875 mmol/L to ULN | 83.3
  At Month 24: >ULN: number analyzed (Participants) | 30
  At Month 24: >ULN | 0
  At Month 30: <1.875 mmol/L: number analyzed (Participants) | 23
  At Month 30: <1.875 mmol/L | 17.4
  At Month 30: 1.875 mmol/L to ULN: number analyzed (Participants) | 23
  At Month 30: 1.875 mmol/L to ULN | 78.3
  At Month 30: >ULN: number analyzed (Participants) | 23
  At Month 30: >ULN | 4.3
  At Month 36: <1.875 mmol/L: number analyzed (Participants) | 1
  At Month 36: <1.875 mmol/L | 0
  At Month 36: 1.875 mmol/L to ULN: number analyzed (Participants) | 1
  At Month 36: 1.875 mmol/L to ULN | 100
  At Month 36: >ULN: number analyzed (Participants) | 1
  At Month 36: >ULN | 0
  At EOT (up to Month 36): <1.875 mmol/L | 13.9
  At EOT (up to Month 36): 1.875 mmol/L to ULN | 83.3
  At EOT (up to Month 36): >ULN | 2.8

9. Secondary Outcome: Change From Baseline (402) in Urinary Calcium Excretion at Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Description: Baseline (402) was defined as the last available pre-dose value in SHP634-402. EOT was defined as the last determination of response during the treatment period (from the date of first dose to the date of last dose + 1 day), was analyzed in addition to the scheduled visits. Here, '0' in the number analyzed field signifies that no participants were evaluable at specified time point.
Time Frame: Baseline (402), At Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Millimole per day (mmol/day)
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 34
Millimole per day (mmol/day)
  Change at Month 6: number analyzed (Participants) | 22
  Change at Month 6 | -0.403 (2.7785)
  Change at Month 12: number analyzed (Participants) | 29
  Change at Month 12 | 0.442 (2.7419)
  Change at Month 18: number analyzed (Participants) | 21
  Change at Month 18 | 0.946 (3.2615)
  Change at Month 24: number analyzed (Participants) | 19
  Change at Month 24 | 1.378 (3.1076)
  Change at Month 30: number analyzed (Participants) | 18
  Change at Month 30 | 2.163 (4.2794)
  Change at Month 36: number analyzed (Participants) | 0
  Change at EOT (up to Month 36) | 1.213 (3.3632)

10. Secondary Outcome: Change From Baseline (402) in Concentration of Serum Phosphate Levels at Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Description: as for outcome 7
Time Frame: Baseline (402), At Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 33
mmol/L
  Change at Month 6: number analyzed (Participants) | 23
  Change at Month 6 | 0.041 (0.2282)
  Change at Month 12: number analyzed (Participants) | 29
  Change at Month 12 | 0.077 (0.2925)
  Change at Month 18: number analyzed (Participants) | 30
  Change at Month 18 | 0.070 (0.3213)
  Change at Month 24: number analyzed (Participants) | 27
  Change at Month 24 | 0.074 (0.2825)
  Change at Month 30: number analyzed (Participants) | 21
  Change at Month 30 | 0.012 (0.2992)
  Change at Month 36: number analyzed (Participants) | 1
  Change at Month 36 | -0.040 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Change at EOT (up to Month 36) | 0.055 (0.2861)

11. Secondary Outcome: Change From Baseline (402) in Calcium Supplement Doses and Elemental Calcium Based on Investigator-prescribed Data and Diary Data at Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Description: as for outcome 7
Time Frame: Baseline, At Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: milligram per day (mg/day)
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 36
milligram per day (mg/day)
  Calcium Prescribed Data: Change at Month 6: number analyzed (Participants) | 24
  Calcium Prescribed Data: Change at Month 6 | 52.1 (547.62)
  Calcium Prescribed Data: Change at Month 12: number analyzed (Participants) | 32
  Calcium Prescribed Data: Change at Month 12 | -125.6 (1189.52)
  Calcium Prescribed Data: Change at Month 18: number analyzed (Participants) | 33
  Calcium Prescribed Data: Change at Month 18 | -150.9 (1140.42)
  Calcium Prescribed Data: Change at Month 24: number analyzed (Participants) | 30
  Calcium Prescribed Data: Change at Month 24 | -146.0 (1401.84)
  Calcium Prescribed Data: Change at Month 30: number analyzed (Participants) | 23
  Calcium Prescribed Data: Change at Month 30 | -105.7 (1262.95)
  Calcium Prescribed Data: Change at Month 36: number analyzed (Participants) | 1
  Calcium Prescribed Data: Change at Month 36 | 230.0 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Calcium Prescribed Data: Change at EOT (up to Month 36) | -237.8 (1208.06)
  Elemental Calcium Prescribed Data: Change at Month 6: number analyzed (Participants) | 24
  Elemental Calcium Prescribed Data: Change at Month 6 | -71.35 (360.730)
  Elemental Calcium Prescribed Data: Change at Month 12: number analyzed (Participants) | 32
  Elemental Calcium Prescribed Data: Change at Month 12 | -201.62 (719.878)
  Elemental Calcium Prescribed Data: Change at Month 18: number analyzed (Participants) | 33
  Elemental Calcium Prescribed Data: Change at Month 18 | -206.40 (727.017)
  Elemental Calcium Prescribed Data: Change at Month 24: number analyzed (Participants) | 30
  Elemental Calcium Prescribed Data: Change at Month 24 | -239.71 (898.529)
  Elemental Calcium Prescribed Data: Change at Month 30: number analyzed (Participants) | 23
  Elemental Calcium Prescribed Data: Change at Month 30 | -175.56 (861.198)
  Elemental Calcium Prescribed Data: Change at Month 36: number analyzed (Participants) | 1
  Elemental Calcium Prescribed Data: Change at Month 36 | -267.70 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Elemental Calcium Prescribed Data: Change at EOT (up to Month 36) | -224.31 (766.956)
  Calcium Diary Data: Change at Month 6: number analyzed (Participants) | 24
  Calcium Diary Data: Change at Month 6 | 537.420 (679.5444)
  Calcium Diary Data: Change at Month 12: number analyzed (Participants) | 32
  Calcium Diary Data: Change at Month 12 | 549.757 (974.4770)
  Calcium Diary Data: Change at Month 18: number analyzed (Participants) | 33
  Calcium Diary Data: Change at Month 18 | 1241.382 (3353.7093)
  Calcium Diary Data: Change at Month 24: number analyzed (Participants) | 30
  Calcium Diary Data: Change at Month 24 | 375.005 (797.0665)
  Calcium Diary Data: Change at Month 30: number analyzed (Participants) | 23
  Calcium Diary Data: Change at Month 30 | 102.174 (240.7955)
  Calcium Diary Data: Change at Month 36: number analyzed (Participants) | 1
  Calcium Diary Data: Change at Month 36 | 0.000 (NA) — Standard deviation could not be calculated because single participant was analyzed
  Calcium Diary Data: Change at EOT (up to Month 36) | 75.545 (220.3270)
  Elemental Calcium Diary Data: Change at Month 6: number analyzed (Participants) | 24
  Elemental Calcium Diary Data: Change at Month 6 | 151.528 (197.2856)
  Elemental Calcium Diary Data: Change at Month 12: number analyzed (Participants) | 32
  Elemental Calcium Diary Data: Change at Month 12 | 194.332 (414.3470)
  Elemental Calcium Diary Data: Change at Month 18: number analyzed (Participants) | 33
  Elemental Calcium Diary Data: Change at Month 18 | 418.160 (1334.7574)
  Elemental Calcium Diary Data: Change at Month 24: number analyzed (Participants) | 30
  Elemental Calcium Diary Data: Change at Month 24 | 145.618 (348.2148)
  Elemental Calcium Diary Data: Change at Month 30: number analyzed (Participants) | 23
  Elemental Calcium Diary Data: Change at Month 30 | 28.854 (67.2635)
  Elemental Calcium Diary Data: Change at Month 36: number analyzed (Participants) | 1
  Elemental Calcium Diary Data: Change at Month 36 | 0.000 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Elemental Calcium Diary Data: Change at EOT (up to Month 36) | 25.868 (80.6473)

12. Secondary Outcome: Change From Baseline (402) in Active Vitamin D Supplement Dose Based on Investigator-prescribed Data and Diary Data at Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Description: as for outcome 7
Time Frame: Baseline (402), At Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: microgram per day (mcg/day)
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 36
microgram per day (mcg/day)
  Prescribed Data: Change at Month 6: number analyzed (Participants) | 24
  Prescribed Data: Change at Month 6 | -0.012 (0.0514)
  Prescribed Data: Change at Month 12: number analyzed (Participants) | 32
  Prescribed Data: Change at Month 12 | -0.056 (0.2747)
  Prescribed Data: Change at Month 18: number analyzed (Participants) | 33
  Prescribed Data: Change at Month 18 | -0.062 (0.3125)
  Prescribed Data: Change at Month 24: number analyzed (Participants) | 30
  Prescribed Data: Change at Month 24 | -0.092 (0.3565)
  Prescribed Data: Change at Month 30: number analyzed (Participants) | 23
  Prescribed Data: Change at Month 30 | -0.034 (0.3559)
  Prescribed Data: Change at Month 36: number analyzed (Participants) | 1
  Prescribed Data: Change at Month 36 | 0.000 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Prescribed Data: Change at EOT (up to Month 36) | -0.063 (0.4022)
  Diary Data: Change at Month 6: number analyzed (Participants) | 24
  Diary Data: Change at Month 6 | 0.063 (0.2117)
  Diary Data: Change at Month 12: number analyzed (Participants) | 32
  Diary Data: Change at Month 12 | 0.032 (0.1109)
  Diary Data: Change at Month 18: number analyzed (Participants) | 33
  Diary Data: Change at Month 18 | 0.015 (0.0606)
  Diary Data: Change at Month 24: number analyzed (Participants) | 30
  Diary Data: Change at Month 24 | 0.092 (0.3742)
  Diary Data: Change at Month 30: number analyzed (Participants) | 23
  Diary Data: Change at Month 30 | 0.000 (0.0000)
  Diary Data: Change at Month 36: number analyzed (Participants) | 1
  Diary Data: Change at Month 36 | 0.000 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Diary Data: Change at EOT (up to Month 36) | 0.000 (0.0000)

13. Secondary Outcome: Change From Baseline (402) in Hypoparathyroidism Symptoms Diary (HPT-SD) at Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Description: The HPT-SD was a 13-item patient-reported outcomes instrument that consists of the following items: symptom subscale (items 1-7), anxiety (item 8), sadness and depression (item 9) and impact subscale (items 10-13). For items 1-9, the individual score ranges from None (0), Mild (1), Moderate (2), Severe (3), Very severe (4) and for items 10-13, it ranges from Not at all (0), somewhat (1), Very much (2). For symptom subscale score was calculated as average score of the items 1-7 and the impact subscale scores was calculated as average score of the items 10-13. The HPT-SD was only collected within the SHP634-402 study, as planned.
Time Frame: Baseline (402), At Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 33
Score on a Scale
  Symptom Subscale: Change at Month 6: number analyzed (Participants) | 22
  Symptom Subscale: Change at Month 6 | 0.06 (0.680)
  Symptom Subscale: Change at Month 12: number analyzed (Participants) | 30
  Symptom Subscale: Change at Month 12 | -0.31 (0.762)
  Symptom Subscale: Change at Month 18: number analyzed (Participants) | 31
  Symptom Subscale: Change at Month 18 | -0.27 (0.831)
  Symptom Subscale: Change at Month 24: number analyzed (Participants) | 27
  Symptom Subscale: Change at Month 24 | -0.25 (0.544)
  Symptom Subscale: Change at Month 30: number analyzed (Participants) | 23
  Symptom Subscale: Change at Month 30 | -0.20 (0.737)
  Symptom Subscale: Change at Month 36: number analyzed (Participants) | 1
  Symptom Subscale: Change at Month 36 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Symptom Subscale: Change at EOT (up to Month 36) | -0.15 (0.867)
  Anxiety: Change at Month 6: number analyzed (Participants) | 22
  Anxiety: Change at Month 6 | 0.1 (0.64)
  Anxiety: Change at Month 12: number analyzed (Participants) | 30
  Anxiety: Change at Month 12 | 0.1 (0.74)
  Anxiety: Change at Month 18: number analyzed (Participants) | 31
  Anxiety: Change at Month 18 | 0.0 (0.68)
  Anxiety: Change at Month 24: number analyzed (Participants) | 27
  Anxiety: Change at Month 24 | 0.1 (0.75)
  Anxiety: Change at Month 30: number analyzed (Participants) | 23
  Anxiety: Change at Month 30 | 0.2 (0.74)
  Anxiety: Change at Month 36: number analyzed (Participants) | 1
  Anxiety: Change at Month 36 | 0.0 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Anxiety: Change at EOT (up to Month 36) | 0.3 (0.80)
  Sadness and Depression: Change at Month 6: number analyzed (Participants) | 22
  Sadness and Depression: Change at Month 6 | 0.3 (0.65)
  Sadness and Depression: Change at Month 12: number analyzed (Participants) | 30
  Sadness and Depression: Change at Month 12 | -0.1 (0.58)
  Sadness and Depression: Change at Month 18: number analyzed (Participants) | 31
  Sadness and Depression: Change at Month 18 | 0.0 (0.66)
  Sadness and Depression: Change at Month 24: number analyzed (Participants) | 27
  Sadness and Depression: Change at Month 24 | 0.3 (0.72)
  Sadness and Depression: Change at Month 30: number analyzed (Participants) | 23
  Sadness and Depression: Change at Month 30 | 0.2 (0.95)
  Sadness and Depression: Change at Month 36: number analyzed (Participants) | 1
  Sadness and Depression: Change at Month 36 | 0.0 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Sadness and Depression: Change at EOT (up to Month 36) | 0.2 (0.95)
  Impact Subscale: Change at Month 6: number analyzed (Participants) | 22
  Impact Subscale: Change at Month 6 | -0.05 (0.391)
  Impact Subscale: Change at Month 12: number analyzed (Participants) | 28
  Impact Subscale: Change at Month 12 | -0.13 (0.400)
  Impact Subscale: Change at Month 18: number analyzed (Participants) | 29
  Impact Subscale: Change at Month 18 | -0.10 (0.363)
  Impact Subscale: Change at Month 24: number analyzed (Participants) | 26
  Impact Subscale: Change at Month 24 | -0.01 (0.335)
  Impact Subscale: Change at Month 30: number analyzed (Participants) | 22
  Impact Subscale: Change at Month 30 | -0.10 (0.413)
  Impact Subscale: Change at Month 36: number analyzed (Participants) | 1
  Impact Subscale: Change at Month 36 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Impact Subscale: Change at EOT (up to Month 36): number analyzed (Participants) | 31
  Impact Subscale: Change at EOT (up to Month 36) | -0.07 (0.377)

14. Secondary Outcome: Change From Baseline (402) in Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) Assessment at Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Description: FACT-Cog assessment was a 37-item tool with each item rated on a 5-point scale ranging from 0 to 4. It included 4 subscales: perceived cognitive impairments (CogPCI) (20 items, Item 1 - 20, score range 0-80), impact of perceived cognitive impairments on quality of life (CogQOL ) (4 items, Item 34 - 37, score range 0-16), comments from others (CogOth) (4 items, Item 21 - 24, score range 0-16) and perceived cognitive ability (CogPCA) (9 items, Item 25 - 33 score range 0-36). CogPCI subscale and comments from others subscale and two others subscale ranged as following: 0 (not at all), 1 (a little bit), 2 (somewhat), 3 (quite a bit) and 4 (very much). For all four subscales of the FACT-cog: higher scores reflect worse cognitive function. Baseline (402): the last available pre-dose value in SHP634-402. EOT: the last determination of response during the treatment period (from the date of first dose to the date of last dose + 1 day), was analyzed in addition to the scheduled visits.
Time Frame: Baseline (402), At Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 36
Score on a Scale
  CogPCI: Change at Month 6: number analyzed (Participants) | 24
  CogPCI: Change at Month 6 | 0.0 (6.88)
  CogPCI: Change at Month 12: number analyzed (Participants) | 33
  CogPCI: Change at Month 12 | 1.0 (9.28)
  CogPCI: Change at Month 18: number analyzed (Participants) | 33
  CogPCI: Change at Month 18 | -1.4 (9.44)
  CogPCI: Change at Month 24: number analyzed (Participants) | 30
  CogPCI: Change at Month 24 | -0.5 (9.35)
  CogPCI: Change at Month 30: number analyzed (Participants) | 26
  CogPCI: Change at Month 30 | -0.3 (10.87)
  CogPCI: Change at Month 36: number analyzed (Participants) | 1
  CogPCI: Change at Month 36 | -1.0 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  CogPCI: Change at EOT (up to Month 36) | -0.4 (11.14)
  CogQOL: Change at Month 6: number analyzed (Participants) | 24
  CogQOL: Change at Month 6 | -0.1 (2.27)
  CogQOL: Change at Month 12: number analyzed (Participants) | 33
  CogQOL: Change at Month 12 | 1.5 (2.92)
  CogQOL: Change at Month 18: number analyzed (Participants) | 33
  CogQOL: Change at Month 18 | 0.2 (3.16)
  CogQOL: Change at Month 24: number analyzed (Participants) | 30
  CogQOL: Change at Month 24 | 1.5 (3.63)
  CogQOL: Change at Month 30: number analyzed (Participants) | 26
  CogQOL: Change at Month 30 | 0.6 (3.20)
  CogQOL: Change at Month 36: number analyzed (Participants) | 1
  CogQOL: Change at Month 36 | 0.0 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  CogQOL: Change at EOT (up to Month 36) | 0.7 (3.20)
  CogOth: Change at Month 6: number analyzed (Participants) | 23
  CogOth: Change at Month 6 | 0.0 (2.10)
  CogOth: Change at Month 12: number analyzed (Participants) | 32
  CogOth: Change at Month 12 | 0.4 (1.85)
  CogOth: Change at Month 18: number analyzed (Participants) | 32
  CogOth: Change at Month 18 | 0.7 (2.46)
  CogOth: Change at Month 24: number analyzed (Participants) | 28
  CogOth: Change at Month 24 | -0.2 (1.89)
  CogOth: Change at Month 30: number analyzed (Participants) | 25
  CogOth: Change at Month 30 | -0.2 (2.79)
  CogOth: Change at Month 36: number analyzed (Participants) | 1
  CogOth: Change at Month 36 | 0.0 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  CogOth: Change at EOT (up to Month 36): number analyzed (Participants) | 35
  CogOth: Change at EOT (up to Month 36) | 0.2 (2.79)
  CogPCA: Change at Month 6: number analyzed (Participants) | 24
  CogPCA: Change at Month 6 | -0.2 (2.60)
  CogPCA: Change at Month 12: number analyzed (Participants) | 33
  CogPCA: Change at Month 12 | -1.1 (5.59)
  CogPCA: Change at Month 18: number analyzed (Participants) | 33
  CogPCA: Change at Month 18 | -0.1 (5.12)
  CogPCA: Change at Month 24: number analyzed (Participants) | 30
  CogPCA: Change at Month 24 | 0.0 (4.41)
  CogPCA: Change at Month 30: number analyzed (Participants) | 26
  CogPCA: Change at Month 30 | 0.2 (6.62)
  CogPCA: Change at Month 36: number analyzed (Participants) | 1
  CogPCA: Change at Month 36 | -2.0 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  CogPCA: Change at EOT (up to Month 36) | 0.3 (4.68)

15. Secondary Outcome: Change From Baseline (402) in Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale Total Score at Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Description: FACIT fatigue questionnaire contains 13 fatigue-related questions. The responses to the 13 items on the FACIT fatigue questionnaire was measured on a 4-point Likert scale (0-4). Thus, the total score ranges from 0 to 52. High scores represent less fatigue and better quality of life. For 2 questions, item 7 'I have energy' and item 8 'I am able to do my usual activities', the item response from questionnaire will be used as item score and no conversion is needed. For the rest of 11 questions, item score was calculated as 4- item response. Fatigue total score was calculated as: Fatigue Total Score = [sum of (item scores)]*13/ (number of items answered). Baseline (402) was defined as the last available pre-dose value in SHP634-402. EOT was defined as the last determination of response during the treatment period (from the date of first dose to the date of last dose + 1 day), was analyzed in addition to the scheduled visits.
Time Frame: Baseline (402), At Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 36
Score on a Scale
  Change at Month 6: number analyzed (Participants) | 24
  Change at Month 6 | -1.41 (4.932)
  Change at Month 12: number analyzed (Participants) | 33
  Change at Month 12 | 0.10 (7.357)
  Change at Month 18: number analyzed (Participants) | 33
  Change at Month 18 | -0.02 (7.467)
  Change at Month 24: number analyzed (Participants) | 30
  Change at Month 24 | -0.13 (8.618)
  Change at Month 30: number analyzed (Participants) | 26
  Change at Month 30 | -1.92 (10.777)
  Change at Month 36: number analyzed (Participants) | 1
  Change at Month 36 | -1.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Change at EOT (up to Month 36) | -1.01 (8.171)

16. Secondary Outcome: Change From Baseline (402) in Hospital Anxiety and Depression Scale (HADS) at Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Description: The HADS was a 14-item scale that generates ordinal data. Seven of the items related to anxiety (Item 1, 3, 5, 7, 9, 11 and 13) and seven related to depression (Item 2, 4, 6, 8, 10, 12 and 14). The scale was designed to avoid reliance on aspects of conditions that are also common somatic symptoms of illness. Each item on the questionnaire was scored from 0-3, therefore, a person can score between 0 and 21 for either anxiety or depression. For each of the two sub-scores, if a participant obtain a score ranged from: 0 to 7, he is considered as "normal"; 8-10 = Borderline abnormal (borderline case) and 11-21 = Abnormal (case). Baseline (402) was defined as the last available pre-dose value in SHP634-402. EOT was defined as the last determination of response during the treatment period (from the date of first dose to the date of last dose + 1 day), was analyzed in addition to the scheduled visits.
Time Frame: Baseline (402), At Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 36
Score on a Scale
  Anxiety Subscale: Change at Month 6: number analyzed (Participants) | 24
  Anxiety Subscale: Change at Month 6 | 0.6 (2.39)
  Anxiety Subscale: Change at Month 12: number analyzed (Participants) | 33
  Anxiety Subscale: Change at Month 12 | -0.5 (2.96)
  Anxiety Subscale: Change at Month 18: number analyzed (Participants) | 33
  Anxiety Subscale: Change at Month 18 | -0.2 (3.74)
  Anxiety Subscale: Change at Month 24: number analyzed (Participants) | 30
  Anxiety Subscale: Change at Month 24 | -1.5 (3.26)
  Anxiety Subscale: Change at Month 30: number analyzed (Participants) | 25
  Anxiety Subscale: Change at Month 30 | -0.4 (3.21)
  Anxiety Subscale: Change at Month 36: number analyzed (Participants) | 1
  Anxiety Subscale: Change at Month 36 | 2.0 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Anxiety Subscale: Change at EOT (up to Month 36) | -0.4 (3.18)
  Depression Subscale: Change at Month 6: number analyzed (Participants) | 24
  Depression Subscale: Change at Month 6 | 0.4 (2.67)
  Depression Subscale: Change at Month 12: number analyzed (Participants) | 33
  Depression Subscale: Change at Month 12 | -0.6 (2.61)
  Depression Subscale: Change at Month 18: number analyzed (Participants) | 33
  Depression Subscale: Change at Month 18 | -0.8 (2.86)
  Depression Subscale: Change at Month 24: number analyzed (Participants) | 30
  Depression Subscale: Change at Month 24 | -0.4 (3.84)
  Depression Subscale: Change at Month 30: number analyzed (Participants) | 25
  Depression Subscale: Change at Month 30 | -1.0 (3.58)
  Depression Subscale: Change at Month 36: number analyzed (Participants) | 1
  Depression Subscale: Change at Month 36 | 1.0 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Depression Subscale: Change at EOT (up to Month 36) | -0.8 (3.35)

17. Secondary Outcome: Change From Baseline (402) in Health-related Quality-of-life Measured With 36-item Short Form Health (SF-36) Survey at Month 12, 24, 36, and EOT (up to Month 36)
Description: SF-36 was a validated questionnaire that questions participants about perceived physical and mental health and function. SF-36 consisted of 8 scaled scores, which were weighted sums of the questions in their section. Each scale was directly transformed into 0-100 scale on the assumption that each question carries equal weight; A score of zero was equivalent to maximum disability and a score of 100 was equivalent to no disability. Eight sections included in SF-36 assessment: vitality (1=none of the time to 5=all of the time), physical functioning (1=yes, limited a lot to 3=no, not limited at all), bodily pain (1=very severe to 6=none), general health (1=poor to 5=excellent), physical role (1=all of the time to 5=none of the time), emotional role (1=all of the time to 5=none of the time), social role (1=all of the time: to 5=none of the time) and mental health (1=all of the time to 5=none of the time). Baseline (402) was defined as the last available pre-dose value in SHP634-402.
Time Frame: Baseline (402), At Month 12, 24, 36, and EOT (up to Month 36)
Population: Safety population consisted of all enrolled participants who received at least 1 dose of rhPTH(1-84) regardless of study (SHP634-402 or AAAE0544 [NCT01199614] core study). Here, overall number of participants analyzed refer to the participants evaluable for this outcome measure and "number analyzed" refer to participants evaluable for this outcome at given categories. Due to the FDA recall, no participant received rhPTH for more than 36 months in the study.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 33
Score on a Scale
  Vitality: Change at Month 12: number analyzed (Participants) | 31
  Vitality: Change at Month 12 | -0.11 (13.485)
  Vitality: Change at Month 24: number analyzed (Participants) | 28
  Vitality: Change at Month 24 | -3.27 (17.641)
  Vitality: Change at Month 36: number analyzed (Participants) | 1
  Vitality: Change at Month 36 | -5.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Vitality: Change at EOT (up to Month 36): number analyzed (Participants) | 32
  Vitality: Change at EOT (up to Month 36) | 0.26 (18.006)
  Physical functioning: Change at Month 12: number analyzed (Participants) | 31
  Physical functioning: Change at Month 12 | 1.61 (14.340)
  Physical functioning: Change at Month 24: number analyzed (Participants) | 28
  Physical functioning: Change at Month 24 | 0.00 (13.676)
  Physical functioning: Change at Month 36: number analyzed (Participants) | 1
  Physical functioning: Change at Month 36 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Physical functioning: Change at EOT (up to Month 36): number analyzed (Participants) | 32
  Physical functioning: Change at EOT (up to Month 36) | 2.66 (20.398)
  Bodily pain: Change at Month 12: number analyzed (Participants) | 31
  Bodily pain: Change at Month 12 | 6.55 (16.287)
  Bodily pain: Change at Month 24: number analyzed (Participants) | 28
  Bodily pain: Change at Month 24 | 3.54 (13.948)
  Bodily pain: Change at Month 36: number analyzed (Participants) | 1
  Bodily pain: Change at Month 36 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Bodily pain: Change at EOT (up to Month 36): number analyzed (Participants) | 32
  Bodily pain: Change at EOT (up to Month 36) | 2.44 (15.546)
  General health: Change at Month 12: number analyzed (Participants) | 32
  General health: Change at Month 12 | 3.28 (12.718)
  General health: Change at Month 24: number analyzed (Participants) | 29
  General health: Change at Month 24 | 0.31 (13.033)
  General health: Change at Month 36: number analyzed (Participants) | 1
  General health: Change at Month 36 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  General health: Change at EOT (up to Month 36) | 0.24 (11.755)
  Physical role: Change at Month 12: number analyzed (Participants) | 31
  Physical role: Change at Month 12 | -1.61 (29.535)
  Physical role: Change at Month 24: number analyzed (Participants) | 28
  Physical role: Change at Month 24 | -6.25 (31.641)
  Physical role: Change at Month 36: number analyzed (Participants) | 1
  Physical role: Change at Month 36 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Physical role: Change at EOT (up to Month 36): number analyzed (Participants) | 32
  Physical role: Change at EOT (up to Month 36) | -5.47 (32.213)
  Emotional role: Change at Month 12: number analyzed (Participants) | 31
  Emotional role: Change at Month 12 | -3.23 (31.453)
  Emotional role: Change at Month 24: number analyzed (Participants) | 28
  Emotional role: Change at Month 24 | -2.38 (40.500)
  Emotional role: Change at Month 36: number analyzed (Participants) | 1
  Emotional role: Change at Month 36 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Emotional role: Change at EOT (up to Month 36): number analyzed (Participants) | 32
  Emotional role: Change at EOT (up to Month 36) | -4.17 (45.398)
  Social role: Change at Month 12: number analyzed (Participants) | 31
  Social role: Change at Month 12 | -3.23 (12.487)
  Social role: Change at Month 24: number analyzed (Participants) | 28
  Social role: Change at Month 24 | -1.79 (19.159)
  Social role: Change at Month 36: number analyzed (Participants) | 1
  Social role: Change at Month 36 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Social role: Change at EOT (up to Month 36): number analyzed (Participants) | 32
  Social role: Change at EOT (up to Month 36) | -1.17 (19.145)
  Mental health: Change at Month 12: number analyzed (Participants) | 31
  Mental health: Change at Month 12 | -0.26 (7.585)
  Mental health: Change at Month 24: number analyzed (Participants) | 28
  Mental health: Change at Month 24 | 1.43 (12.845)
  Mental health: Change at Month 36: number analyzed (Participants) | 1
  Mental health: Change at Month 36 | 4.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Mental health: Change at EOT (up to Month 36): number analyzed (Participants) | 32
  Mental health: Change at EOT (up to Month 36) | 0.50 (12.801)

18. Secondary Outcome: Change From Baseline (402) in Concentration of Bone Turnover Markers at Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Description: Change from baseline in concentration of bone turnover markers included; Serum carboxy-terminal 4 telopeptide of type I collagen [s-CTX], procollagen type I amino-terminal propeptide [P1NP], osteocalcin, and sclerostin. Baseline (402) was defined as the last available pre-dose value in SHP634-402. EOT was defined as the last determination of response during the treatment period (from the date of first dose to the date of last dose + 1 day), was analyzed in addition to the scheduled visits. Here, '0' in the number analyzed field signifies that no participants were evaluable at specified time point.
Time Frame: Baseline (402), At Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 15
mcg/L
  s-CTX: Change at Month 6: number analyzed (Participants) | 7
  s-CTX: Change at Month 6 | -0.082 (0.1053)
  s-CTX: Change at Month 12: number analyzed (Participants) | 8
  s-CTX: Change at Month 12 | -0.190 (0.9847)
  s-CTX: Change at Month 18: number analyzed (Participants) | 10
  s-CTX: Change at Month 18 | 0.036 (0.3030)
  s-CTX: Change at Month 24: number analyzed (Participants) | 8
  s-CTX: Change at Month 24 | 0.201 (0.3985)
  s-CTX: Change at Month 30: number analyzed (Participants) | 5
  s-CTX: Change at Month 30 | -0.204 (0.2896)
  s-CTX: Change at Month 36: number analyzed (Participants) | 0
  s-CTX: Change at EOT (up to Month 36): number analyzed (Participants) | 11
  s-CTX: Change at EOT (up to Month 36) | -0.136 (0.5429)
  P1NP: Change at Month 6: number analyzed (Participants) | 11
  P1NP: Change at Month 6 | -3.12 (30.262)
  P1NP: Change at Month 12: number analyzed (Participants) | 13
  P1NP: Change at Month 12 | 33.94 (55.080)
  P1NP: Change at Month 18: number analyzed (Participants) | 14
  P1NP: Change at Month 18 | 31.06 (137.665)
  P1NP: Change at Month 24: number analyzed (Participants) | 11
  P1NP: Change at Month 24 | 37.09 (152.162)
  P1NP: Change at Month 30: number analyzed (Participants) | 8
  P1NP: Change at Month 30 | 30.95 (85.345)
  P1NP: Change at Month 36: number analyzed (Participants) | 0
  P1NP: Change at EOT (up to Month 36) | 80.90 (175.466)
  Osteocalcin: Change at Month 6: number analyzed (Participants) | 9
  Osteocalcin: Change at Month 6 | -4.020 (11.6418)
  Osteocalcin: Change at Month 12: number analyzed (Participants) | 11
  Osteocalcin: Change at Month 12 | -1.199 (44.2510)
  Osteocalcin: Change at Month 18: number analyzed (Participants) | 12
  Osteocalcin: Change at Month 18 | -0.310 (43.7374)
  Osteocalcin: Change at Month 24: number analyzed (Participants) | 10
  Osteocalcin: Change at Month 24 | 23.483 (31.7005)
  Osteocalcin: Change at Month 30: number analyzed (Participants) | 7
  Osteocalcin: Change at Month 30 | 3.674 (36.8616)
  Osteocalcin: Change at Month 36: number analyzed (Participants) | 0
  Osteocalcin: Change at EOT (up to Month 36): number analyzed (Participants) | 13
  Osteocalcin: Change at EOT (up to Month 36) | 29.232 (65.9276)
  Sclerostin: Change at Month 6: number analyzed (Participants) | 11
  Sclerostin: Change at Month 6 | 0.013 (0.1678)
  Sclerostin: Change at Month 12: number analyzed (Participants) | 13
  Sclerostin: Change at Month 12 | 0.071 (0.1657)
  Sclerostin: Change at Month 18: number analyzed (Participants) | 14
  Sclerostin: Change at Month 18 | 0.097 (0.2512)
  Sclerostin: Change at Month 24: number analyzed (Participants) | 11
  Sclerostin: Change at Month 24 | 0.092 (0.1978)
  Sclerostin: Change at Month 30: number analyzed (Participants) | 8
  Sclerostin: Change at Month 30 | 0.029 (0.1302)
  Sclerostin: Change at Month 36: number analyzed (Participants) | 0
  Sclerostin: Change at EOT (up to Month 36) | 0.075 (0.1651)

19. Secondary Outcome: Change From Baseline (402) in Concentration of Bone Turnover Marker for Bone Specific Alkaline Phosphatase and Tartrate-resistant Acid Phosphatase-5b at Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Description: Change from baseline in concentration of bone turnover markers included, bone specific alkaline phosphatase [BSAP] and tartrate-resistant acid phosphatase-5b (TRAP-5b). Baseline (402) was defined as the last available pre-dose value in SHP634-402. EOT was defined as the last determination of response during the treatment period (from the date of first dose to the date of last dose + 1 day), was analyzed in addition to the scheduled visits. Here, '0' in the number analyzed field signifies that no participants were evaluable at specified time point.
Time Frame: Baseline (402), At Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 15
Units per liter (U/L)
  BSAP: Change at Month 6: number analyzed (Participants) | 11
  BSAP: Change at Month 6 | -1.194 (4.8791)
  BSAP: Change at Month 12: number analyzed (Participants) | 13
  BSAP: Change at Month 12 | 4.310 (11.8965)
  BSAP: Change at Month 18: number analyzed (Participants) | 14
  BSAP: Change at Month 18 | 4.824 (13.0980)
  BSAP: Change at Month 24: number analyzed (Participants) | 11
  BSAP: Change at Month 24 | 11.546 (14.1455)
  BSAP: Change at Month 30: number analyzed (Participants) | 8
  BSAP: Change at Month 30 | 2.124 (9.6951)
  BSAP: Change at Month 36: number analyzed (Participants) | 0
  BSAP: Change at EOT (up to Month 36) | 7.167 (12.4372)
  TRAP-5b: Change at Month 6: number analyzed (Participants) | 11
  TRAP-5b: Change at Month 6 | -0.236 (0.7336)
  TRAP-5b: Change at Month 12: number analyzed (Participants) | 13
  TRAP-5b: Change at Month 12 | 0.946 (1.8702)
  TRAP-5b: Change at Month 18: number analyzed (Participants) | 14
  TRAP-5b: Change at Month 18 | 1.798 (4.3422)
  TRAP-5b: Change at Month 24: number analyzed (Participants) | 11
  TRAP-5b: Change at Month 24 | 2.347 (2.3850)
  TRAP-5b: Change at Month 30: number analyzed (Participants) | 8
  TRAP-5b: Change at Month 30 | 1.254 (4.2890)
  TRAP-5b: Change at Month 36: number analyzed (Participants) | 0
  TRAP-5b: Change at EOT (up to Month 36) | 1.336 (3.2241)

20. Secondary Outcome: Change From Baseline (402) in Bone Architecture Evaluated Using Dual-energy X-ray Absorptiometry (DXA) for Bone Mineral Density (BMD) at Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Description: Change from baseline in bone architecture was assessed by using DXA. The DXA scans was evaluated for BMD of the lumbar spine (vertebra L1, L2, L3, L4), total hip and femoral neck, and distal radius. Baseline (402) was defined as the last available pre-dose value in SHP634-402. EOT was defined as the last determination of response during the treatment period (from the date of first dose to the date of last dose + 1 day), was analyzed in addition to the scheduled visits. Here, '0' in the number analyzed field signifies that no participants were evaluable at specified time point.
Time Frame: Baseline, At Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Grams per square centimeter (g/cm^2)
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 24
Grams per square centimeter (g/cm^2)
  Lumbar Spine Total: Change at Month 6: number analyzed (Participants) | 17
  Lumbar Spine Total: Change at Month 6 | -0.027 (0.0386)
  Lumbar Spine Total: Change at Month 12: number analyzed (Participants) | 23
  Lumbar Spine Total: Change at Month 12 | -0.020 (0.0398)
  Lumbar Spine Total: Change at Month 18: number analyzed (Participants) | 22
  Lumbar Spine Total: Change at Month 18 | -0.012 (0.0385)
  Lumbar Spine Total: Change at Month 24: number analyzed (Participants) | 18
  Lumbar Spine Total: Change at Month 24 | -0.008 (0.0545)
  Lumbar Spine Total: Change at Month 30: number analyzed (Participants) | 16
  Lumbar Spine Total: Change at Month 30 | -0.021 (0.0549)
  Lumbar Spine Total: Change at Month 36: number analyzed (Participants) | 0
  Lumbar Spine Total: Change at EOT (up to Month 36) | -0.024 (0.0524)
  Lumbar L1: Change at Month 6: number analyzed (Participants) | 14
  Lumbar L1: Change at Month 6 | 0.000 (0.0334)
  Lumbar L1: Change at Month 12: number analyzed (Participants) | 19
  Lumbar L1: Change at Month 12 | 0.001 (0.0374)
  Lumbar L1: Change at Month 18: number analyzed (Participants) | 18
  Lumbar L1: Change at Month 18 | 0.003 (0.0426)
  Lumbar L1: Change at Month 24: number analyzed (Participants) | 15
  Lumbar L1: Change at Month 24 | 0.018 (0.0552)
  Lumbar L1: Change at Month 30: number analyzed (Participants) | 13
  Lumbar L1: Change at Month 30 | -0.006 (0.0656)
  Lumbar L1: Change at Month 36: number analyzed (Participants) | 0
  Lumbar L1: Change at EOT (up to Month 36): number analyzed (Participants) | 20
  Lumbar L1: Change at EOT (up to Month 36) | 0.005 (0.0641)
  Lumbar L2: Change at Month 6: number analyzed (Participants) | 15
  Lumbar L2: Change at Month 6 | -0.020 (0.0276)
  Lumbar L2: Change at Month 12: number analyzed (Participants) | 20
  Lumbar L2: Change at Month 12 | -0.017 (0.0399)
  Lumbar L2: Change at Month 18: number analyzed (Participants) | 20
  Lumbar L2: Change at Month 18 | -0.006 (0.0428)
  Lumbar L2: Change at Month 24: number analyzed (Participants) | 16
  Lumbar L2: Change at Month 24 | -0.001 (0.0518)
  Lumbar L2: Change at Month 30: number analyzed (Participants) | 13
  Lumbar L2: Change at Month 30 | -0.012 (0.0560)
  Lumbar L2: Change at Month 36: number analyzed (Participants) | 0
  Lumbar L2: Change at EOT (up to Month 36): number analyzed (Participants) | 21
  Lumbar L2: Change at EOT (up to Month 36) | -0.018 (0.0487)
  Lumbar L3: Change at Month 6: number analyzed (Participants) | 15
  Lumbar L3: Change at Month 6 | -0.018 (0.0325)
  Lumbar L3: Change at Month 12: number analyzed (Participants) | 21
  Lumbar L3: Change at Month 12 | -0.015 (0.0466)
  Lumbar L3: Change at Month 18: number analyzed (Participants) | 21
  Lumbar L3: Change at Month 18 | -0.012 (0.0538)
  Lumbar L3: Change at Month 24: number analyzed (Participants) | 16
  Lumbar L3: Change at Month 24 | -0.001 (0.0495)
  Lumbar L3: Change at Month 30: number analyzed (Participants) | 14
  Lumbar L3: Change at Month 30 | -0.013 (0.0478)
  Lumbar L3: Change at Month 36: number analyzed (Participants) | 0
  Lumbar L3: Change at EOT (up to Month 36): number analyzed (Participants) | 22
  Lumbar L3: Change at EOT (up to Month 36) | -0.016 (0.0541)
  Lumbar L4: Change at Month 6: number analyzed (Participants) | 14
  Lumbar L4: Change at Month 6 | -0.015 (0.0328)
  Lumbar L4: Change at Month 12: number analyzed (Participants) | 19
  Lumbar L4: Change at Month 12 | -0.010 (0.0362)
  Lumbar L4: Change at Month 18: number analyzed (Participants) | 19
  Lumbar L4: Change at Month 18 | -0.013 (0.0319)
  Lumbar L4: Change at Month 24: number analyzed (Participants) | 16
  Lumbar L4: Change at Month 24 | -0.004 (0.0546)
  Lumbar L4: Change at Month 30: number analyzed (Participants) | 15
  Lumbar L4: Change at Month 30 | -0.014 (0.0513)
  Lumbar L4: Change at Month 36: number analyzed (Participants) | 0
  Lumbar L4: Change at EOT (up to Month 36): number analyzed (Participants) | 21
  Lumbar L4: Change at EOT (up to Month 36) | -0.023 (0.0497)
  Femoral Neck: Change at Month 6: number analyzed (Participants) | 17
  Femoral Neck: Change at Month 6 | -0.010 (0.0468)
  Femoral Neck: Change at Month 12: number analyzed (Participants) | 23
  Femoral Neck: Change at Month 12 | -0.027 (0.0470)
  Femoral Neck: Change at Month 18: number analyzed (Participants) | 22
  Femoral Neck: Change at Month 18 | -0.025 (0.0543)
  Femoral Neck: Change at Month 24: number analyzed (Participants) | 18
  Femoral Neck: Change at Month 24 | -0.032 (0.0574)
  Femoral Neck: Change at Month 30: number analyzed (Participants) | 16
  Femoral Neck: Change at Month 30 | -0.020 (0.0483)
  Femoral Neck: Change at Month 36: number analyzed (Participants) | 0
  Femoral Neck: Change at EOT (up to Month 36) | -0.018 (0.0467)
  Total Hip: Change at Month 6: number analyzed (Participants) | 17
  Total Hip: Change at Month 6 | -0.005 (0.0213)
  Total Hip: Change at Month 12: number analyzed (Participants) | 23
  Total Hip: Change at Month 12 | -0.004 (0.0224)
  Total Hip: Change at Month 18: number analyzed (Participants) | 22
  Total Hip: Change at Month 18 | -0.001 (0.0293)
  Total Hip: Change at Month 24: number analyzed (Participants) | 18
  Total Hip: Change at Month 24 | -0.008 (0.0299)
  Total Hip: Change at Month 30: number analyzed (Participants) | 16
  Total Hip: Change at Month 30 | -0.003 (0.0359)
  Total Hip: Change at Month 36: number analyzed (Participants) | 0
  Total Hip: Change at EOT (up to Month 36) | -0.013 (0.0358)
  Distal Radius: Change at Month 6: number analyzed (Participants) | 17
  Distal Radius: Change at Month 6 | 0.032 (0.1204)
  Distal Radius: Change at Month 12: number analyzed (Participants) | 23
  Distal Radius: Change at Month 12 | 0.018 (0.1104)
  Distal Radius: Change at Month 18: number analyzed (Participants) | 22
  Distal Radius: Change at Month 18 | 0.020 (0.1193)
  Distal Radius: Change at Month 24: number analyzed (Participants) | 18
  Distal Radius: Change at Month 24 | 0.024 (0.1278)
  Distal Radius: Change at Month 30: number analyzed (Participants) | 16
  Distal Radius: Change at Month 30 | 0.024 (0.1276)
  Distal Radius: Change at Month 36: number analyzed (Participants) | 0
  Distal Radius: Change at EOT (up to Month 36) | 0.011 (0.1049)

21. Secondary Outcome: Change From Baseline (402) in Bone Architecture Evaluated Using Dual-energy X-ray Absorptiometry (DXA) for Total T-scores at Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Description: Change from baseline in bone architecture was assessed by using DXA. The DXA scans was evaluated for Total T-score of the lumbar spine (vertebra L1-L4), hip (total and femoral neck), and ⅓ distal radius. Baseline (402) was defined as the last available pre-dose value in SHP634-402. The T-score was a comparison of a person's bone density with that of a healthy 30-year-old adult of the same sex and ethnicity. T-score included: Normal: >= -1; Osteopenia: < -1 and > -2.5; Osteoporosis: <= -2.5. A lower T-score implies a lower bone mineral density. EOT was defined as the last determination of response during the treatment period (from the date of first dose to the date of last dose + 1 day), was analyzed in addition to the scheduled visits. Here, '0' in the number analyzed field signifies that no participants were evaluable at specified time point.
Time Frame: Baseline, At Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 24
T-score
  Lumbar Spine Total: Change at Month 6: number analyzed (Participants) | 17
  Lumbar Spine Total: Change at Month 6 | -0.16 (0.343)
  Lumbar Spine Total: Change at Month 12: number analyzed (Participants) | 23
  Lumbar Spine Total: Change at Month 12 | -0.12 (0.331)
  Lumbar Spine Total: Change at Month 18: number analyzed (Participants) | 22
  Lumbar Spine Total: Change at Month 18 | -0.09 (0.338)
  Lumbar Spine Total: Change at Month 24: number analyzed (Participants) | 18
  Lumbar Spine Total: Change at Month 24 | -0.04 (0.477)
  Lumbar Spine Total: Change at Month 30: number analyzed (Participants) | 16
  Lumbar Spine Total: Change at Month 30 | -0.16 (0.506)
  Lumbar Spine Total: Change at Month 36: number analyzed (Participants) | 0
  Lumbar Spine Total: Change at EOT (up to Month 36) | -0.18 (0.476)
  Lumbar Spine L1: Change at Month 6: number analyzed (Participants) | 14
  Lumbar Spine L1: Change at Month 6 | -0.01 (0.293)
  Lumbar Spine L1: Change at Month 12: number analyzed (Participants) | 19
  Lumbar Spine L1: Change at Month 12 | 0.01 (0.346)
  Lumbar Spine L1: Change at Month 18: number analyzed (Participants) | 18
  Lumbar Spine L1: Change at Month 18 | 0.01 (0.394)
  Lumbar Spine L1: Change at Month 24: number analyzed (Participants) | 15
  Lumbar Spine L1: Change at Month 24 | 0.16 (0.508)
  Lumbar Spine L1: Change at Month 30: number analyzed (Participants) | 13
  Lumbar Spine L1: Change at Month 30 | -0.05 (0.598)
  Lumbar Spine L1: Change at Month 36: number analyzed (Participants) | 0
  Lumbar Spine L1: Change at Month EOT (up to Month 36): number analyzed (Participants) | 20
  Lumbar Spine L1: Change at Month EOT (up to Month 36) | 0.04 (0.588)
  Lumbar Spine L2: Change at Month 6: number analyzed (Participants) | 15
  Lumbar Spine L2: Change at Month 6 | -0.17 (0.243)
  Lumbar Spine L2: Change at Month 12: number analyzed (Participants) | 20
  Lumbar Spine L2: Change at Month 12 | -0.15 (0.361)
  Lumbar Spine L2: Change at Month 18: number analyzed (Participants) | 20
  Lumbar Spine L2: Change at Month 18 | -0.05 (0.394)
  Lumbar Spine L2: Change at Month 24: number analyzed (Participants) | 16
  Lumbar Spine L2: Change at Month 24 | 0.01 (0.477)
  Lumbar Spine L2: Change at Month 30: number analyzed (Participants) | 13
  Lumbar Spine L2: Change at Month 30 | -0.10 (0.512)
  Lumbar Spine L2: Change at Month 36: number analyzed (Participants) | 0
  Lumbar Spine L2: Change at EOT (up to Month 36): number analyzed (Participants) | 21
  Lumbar Spine L2: Change at EOT (up to Month 36) | -0.15 (0.440)
  Lumbar Spine L3: Change at Month 6: number analyzed (Participants) | 15
  Lumbar Spine L3: Change at Month 6 | -0.16 (0.304)
  Lumbar Spine L3: Change at Month 12: number analyzed (Participants) | 21
  Lumbar Spine L3: Change at Month 12 | -0.12 (0.424)
  Lumbar Spine L3: Change at Month 18: number analyzed (Participants) | 21
  Lumbar Spine L3: Change at Month 18 | -0.10 (0.518)
  Lumbar Spine L3: Change at Month 24: number analyzed (Participants) | 16
  Lumbar Spine L3: Change at Month 24 | 0.03 (0.468)
  Lumbar Spine L3: Change at Month 30: number analyzed (Participants) | 14
  Lumbar Spine L3: Change at Month 30 | -0.11 (0.461)
  Lumbar Spine L3: Change at Month 36: number analyzed (Participants) | 0
  Lumbar Spine L3: Change at EOT (up to Month 36): number analyzed (Participants) | 22
  Lumbar Spine L3: Change at EOT (up to Month 36) | -0.14 (0.509)
  Lumbar Spine L4: Change at Month 6: number analyzed (Participants) | 14
  Lumbar Spine L4: Change at Month 6 | -0.13 (0.287)
  Lumbar Spine L4: Change at Month 12: number analyzed (Participants) | 19
  Lumbar Spine L4: Change at Month 12 | -0.09 (0.336)
  Lumbar Spine L4: Change at Month 18: number analyzed (Participants) | 19
  Lumbar Spine L4: Change at Month 18 | -0.12 (0.306)
  Lumbar Spine L4: Change at Month 24: number analyzed (Participants) | 16
  Lumbar Spine L4: Change at Month 24 | -0.04 (0.484)
  Lumbar Spine L4: Change at Month 30: number analyzed (Participants) | 15
  Lumbar Spine L4: Change at Month 30 | -0.14 (0.479)
  Lumbar Spine L4: Change at Month 36: number analyzed (Participants) | 0
  Lumbar Spine L4: Change at EOT (up to Month 36): number analyzed (Participants) | 21
  Lumbar Spine L4: Change at EOT (up to Month 36) | -0.21 (0.456)
  Femoral Neck: Change at Month 6: number analyzed (Participants) | 17
  Femoral Neck: Change at Month 6 | -0.06 (0.386)
  Femoral Neck: Change at Month 12: number analyzed (Participants) | 23
  Femoral Neck: Change at Month 12 | -0.21 (0.390)
  Femoral Neck: Change at Month 18: number analyzed (Participants) | 22
  Femoral Neck: Change at Month 18 | -0.21 (0.448)
  Femoral Neck: Change at Month 24: number analyzed (Participants) | 18
  Femoral Neck: Change at Month 24 | -0.26 (0.462)
  Femoral Neck: Change at Month 30: number analyzed (Participants) | 16
  Femoral Neck: Change at Month 30 | -0.17 (0.451)
  Femoral Neck: Change at Month 36: number analyzed (Participants) | 0
  Femoral Neck: Change at EOT (up to Month 36) | -0.16 (0.427)
  Total Hip: Change at Month 6: number analyzed (Participants) | 17
  Total Hip: Change at Month 6 | -0.02 (0.194)
  Total Hip: Change at Month 12: number analyzed (Participants) | 23
  Total Hip: Change at Month 12 | -0.03 (0.200)
  Total Hip: Change at Month 18: number analyzed (Participants) | 22
  Total Hip: Change at Month 18 | 0.00 (0.240)
  Total Hip: Change at Month 24: number analyzed (Participants) | 18
  Total Hip: Change at Month 24 | -0.07 (0.274)
  Total Hip: Change at Month 30: number analyzed (Participants) | 16
  Total Hip: Change at Month 30 | -0.02 (0.306)
  Total Hip: Change at Month 36: number analyzed (Participants) | 0
  Total Hip: Change at EOT (up to Month 36) | -0.10 (0.304)
  Distal 1/3 Radius: Change at Month 6: number analyzed (Participants) | 17
  Distal 1/3 Radius: Change at Month 6 | 0.00 (0.408)
  Distal 1/3 Radius: Change at Month 12: number analyzed (Participants) | 23
  Distal 1/3 Radius: Change at Month 12 | -0.09 (0.332)
  Distal 1/3 Radius: Change at Month 18: number analyzed (Participants) | 22
  Distal 1/3 Radius: Change at Month 18 | -0.07 (0.385)
  Distal 1/3 Radius: Change at Month 24: number analyzed (Participants) | 18
  Distal 1/3 Radius: Change at Month 24 | -0.11 (0.342)
  Distal 1/3 Radius: Change at Month 30: number analyzed (Participants) | 16
  Distal 1/3 Radius: Change at Month 30 | -0.16 (0.462)
  Distal 1/3 Radius: Change at Month 36: number analyzed (Participants) | 0
  Distal 1/3 Radius: Change at EOT (up to Month 36) | -0.22 (0.359)

22. Secondary Outcome: Change From Baseline (402) in Bone Architecture Evaluated Using High-resolution Peripheral Quantitative Computerized Tomography (HRpQCT) for Total Area of Radius and Tibia at Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Description: Change from baseline in bone architecture was assessed by using HRpQCT. The HRpQCT analyses included both radius and tibia of total area position. Baseline (402) was defined as the last available pre-dose value in SHP634-402. EOT was defined as the last determination of response during the treatment period (from the date of first dose to the date of last dose + 1 day), was analyzed in addition to the scheduled visits. Here, '0' in the number analyzed field signifies that no participants were evaluable at specified time point.
Time Frame: Baseline (402), At Month 6, 12, 18, 24, 30, 36, and EOT (up to Month 36)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Millimeter square (mm^2)
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 28
Millimeter square (mm^2)
  Total Area Position: Radius, Change at Month 6: number analyzed (Participants) | 18
  Total Area Position: Radius, Change at Month 6 | -2.99 (12.143)
  Total Area Position: Radius, Change at Month 12: number analyzed (Participants) | 19
  Total Area Position: Radius, Change at Month 12 | -1.36 (9.358)
  Total Area Position: Radius, Change at Month 18: number analyzed (Participants) | 24
  Total Area Position: Radius, Change at Month 18 | -3.59 (12.111)
  Total Area Position: Radius, Change at Month 24: number analyzed (Participants) | 20
  Total Area Position: Radius, Change at Month 24 | -5.31 (13.761)
  Total Area Position: Radius, Change at Month 30: number analyzed (Participants) | 18
  Total Area Position: Radius, Change at Month 30 | -6.64 (15.009)
  Total Area Position: Radius, Change at Month 36: number analyzed (Participants) | 0
  Total Area Position: Radius, Change at EOT (up to Month 36): number analyzed (Participants) | 27
  Total Area Position: Radius, Change at EOT (up to Month 36) | -2.21 (13.908)
  Total Area Position: Tibia, Change at Month 6: number analyzed (Participants) | 16
  Total Area Position: Tibia, Change at Month 6 | -5.34 (20.594)
  Total Area Position: Tibia, Change at Month 12: number analyzed (Participants) | 20
  Total Area Position: Tibia, Change at Month 12 | -2.10 (2.941)
  Total Area Position: Tibia, Change at Month 18: number analyzed (Participants) | 24
  Total Area Position: Tibia, Change at Month 18 | -6.02 (16.858)
  Total Area Position: Tibia, Change at Month 24: number analyzed (Participants) | 21
  Total Area Position: Tibia, Change at Month 24 | -6.71 (17.861)
  Total Area Position: Tibia, Change at Month 30: number analyzed (Participants) | 19
  Total Area Position: Tibia, Change at Month 30 | -0.93 (6.703)
  Total Area Position: Tibia, Change at Month 36: number analyzed (Participants) | 0
  Total Area Position: Tibia, Change at EOT (up to Month 36) | -1.21 (6.391)

23. Secondary Outcome: Mean Bone Histology (Biopsy) of Adjusted Apposition Rate and Cancellous Minimum Apposition Rate at Month 12, and EOT (up to Month 36)
Description: Bone histology parameters consisted of adjusted apposition rate and cancellous minimum apposition rate. An optional transiliac bone biopsy was performed for willing participants, at the discretion of the investigator a maximum of three time. EOT was defined as the last determination of response during the treatment period (from the date of first dose to the date of last dose + 1 day), was analyzed in addition to the scheduled visits.
Time Frame: At Month 12, and EOT (up to Month 36)
Population: Safety population consisted of all enrolled participants who received at least dose of rhPTH(1-84) regardless of study (SHP634-402 or AAAE0544 [NCT01199614] core study). Here, overall number of participants analyzed refer to the participants evaluable for this outcome measure and "number analyzed" refer to participants evaluable for this outcome at given categories. Due to the FDA recall, no participant received rhPTH for more than 36 months in the study.
Measure: Mean (Standard Deviation); unit: Micrometer per day (mcm/d)
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 4
Micrometer per day (mcm/d)
  Adjusted Apposition rate: At Month 12: number analyzed (Participants) | 3
  Adjusted Apposition rate: At Month 12 | 0.207 (0.2043)
  Adjusted Apposition rate: At EOT (up to Month 36) | 0.273 (0.2125)
  Cancellous Min Apposition Rate: At Month 12: number analyzed (Participants) | 3
  Cancellous Min Apposition Rate: At Month 12 | 0.453 (0.1604)
  Cancellous Min Apposition Rate: At EOT (up to Month 36) | 0.485 (0.1455)

24. Secondary Outcome: Mean Bone Histology (Biopsy) of Bone Formation Rate at Month 12, and EOT (up to Month 36)
Description: Bone histology parameters consisted of bone formation rate. An optional transiliac bone biopsy was performed for willing participants, at the discretion of the investigator a maximum of three time. EOT was defined as the last determination of response during the treatment period (from the date of first dose to the date of last dose + 1 day), was analyzed in addition to the scheduled visits. Here, "mcm^3/mcm^2/d" is abbreviated as micro cubic meter per micro square meter per day.
Time Frame: At Month 12, and EOT (up to Month 36)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mcm^3/mcm^2/d
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 4
mcm^3/mcm^2/d
  Bone Formation Rate: At Month 12: number analyzed (Participants) | 3
  Bone Formation Rate: At Month 12 | 0.0360 (0.04233)
  Bone Formation Rate: At EOT (up to Month 36) | 0.0665 (0.07011)

25. Secondary Outcome: Mean Bone Histology (Biopsy) of Cancellous Bone Volume, Cancellous Eroded Surface, Cancellous Mineral Surface, And Cancellous Osteoid Surface at Month 12, and EOT (up to Month 36)
Description: Bone histology parameters consisted of cancellous bone volume, cancellous eroded surface, cancellous mineral surface, and cancellous osteoid surface. An optional transiliac bone biopsy was performed for willing participants, at the discretion of the investigator a maximum of three time. EOT was defined as the last determination of response during the treatment period (from the date of first dose to the date of last dose + 1 day), was analyzed in addition to the scheduled visits.
Time Frame: At Month 12, and EOT (up to Month 36)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Percentage of bone histology
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 4
Percentage of bone histology
  Cancellous Bone Volume: At Month 12: number analyzed (Participants) | 3
  Cancellous Bone Volume: At Month 12 | 32.863 (9.3280)
  Cancellous Bone Volume: At EOT (up to Month 36) | 34.988 (8.7210)
  Cancellous Eroded Surface: At Month 12: number analyzed (Participants) | 3
  Cancellous Eroded Surface: At Month 12 | 10.373 (5.1763)
  Cancellous Eroded Surface: At EOT (up to Month 36) | 12.575 (6.1034)
  Cancellous Mineral Surface: At Month 12: number analyzed (Participants) | 3
  Cancellous Mineral Surface: At Month 12 | 6.973 (6.3212)
  Cancellous Mineral Surface: At EOT (up to Month 36) | 12.028 (11.3497)
  Cancellous Osteoid Surface: At Month 12: number analyzed (Participants) | 3
  Cancellous Osteoid Surface: At Month 12 | 17.863 (14.2300)
  Cancellous Osteoid Surface: At EOT (up to Month 36) | 21.803 (14.0379)

26. Secondary Outcome: Mean Bone Histology (Biopsy) of Cancellous Osteoid Thickness and Cortical Width at Month 12, and EOT (up to Month 36)
Description: Bone histology parameters consisted of cancellous osteoid thickness and cortical width. An optional transiliac bone biopsy was performed for willing participants, at the discretion of the investigator a maximum of three time. EOT was defined as the last determination of response during the treatment period (from the date of first dose to the date of last dose + 1 day), was analyzed in addition to the scheduled visits.
Time Frame: At Month 12, and EOT (up to Month 36)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Micrometer (mcm)
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 4
Micrometer (mcm)
  Cancellous Osteoid Thickness: At Month 12: number analyzed (Participants) | 3
  Cancellous Osteoid Thickness: At Month 12 | 6.667 (2.9913)
  Cancellous Osteoid Thickness: At EOT (up to Month 36): number analyzed (Participants) | 3
  Cancellous Osteoid Thickness: At EOT (up to Month 36) | 6.667 (2.9913)
  Cortical Width: At Month 12: number analyzed (Participants) | 3
  Cortical Width: At Month 12 | 668.677 (277.1239)
  Cortical Width: At EOT (up to Month 36) | 698.913 (234.2120)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to end of study (up to 38 months)
Arm/Group | rhPTH(1-84)
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 6/39
Other Adverse Events (participants affected / at risk) | 34/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhPTH(1-84) (N=39)
Angina pectoris (Cardiac disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Hypobarism (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhPTH(1-84) (N=39)
Hypothyroidism (Endocrine disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (5)
Drug hypersensitivity (Immune system disorders) | 2 (2)
Seasonal allergy (Immune system disorders) | 2 (2)
Bronchitis (Infections and infestations) | 3 (4)
Influenza (Infections and infestations) | 5 (5)
Nasopharyngitis (Infections and infestations) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 5 (6)
Pneumonia (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Tooth infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 5 (5)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2)
Ligament rupture (Injury, poisoning and procedural complications) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 10 (17)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 16 (17)
Depression (Psychiatric disorders) | 8 (8)
Insomnia (Psychiatric disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 6 (7)
Varicose vein (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (4):
  • Study Protocol: Original (2016-05-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT02910466/Prot_000.pdf
  • Study Protocol: Amendment 1 (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT02910466/Prot_001.pdf
  • Study Protocol: Amendment 2 (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT02910466/Prot_002.pdf
  • Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/66/NCT02910466/SAP_003.pdf